CLINICAL TRIAL: NCT00780403
Title: A Multi-Center, Pediatric, Open-Label, Preference Study of Desloratadine 2.5 mg Reditab (SCH34117) and Zyrtec ® 5.0 mg Chewable Tablet Medications
Brief Title: Multi-Center, Pediatric, Open-Label, Preference Study of Desloratadine 2.5 mg Reditab (SCH34117) and Zyrtec ® 5.0 mg Chewable Tablet Medications (Study P04573) (Completed)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: P04573
Record Dates: First submitted 2008-10-23; First posted 2008-10-27 (Estimated); Results first posted 2010-07-30 (Estimated); Last update posted 2022-02-09 (Actual); Status verified 2022-02

CONDITIONS: Allergies
MeSH Terms: conditions — Hypersensitivity | interventions — desloratadine; Cetirizine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- RediTab/Zyrtec (Active Comparator): Subjects received a single dose of desloratadine RediTab followed 8-10 minutes later by a single dose of Zyrtec chewable tablet followed thereafter by a statement of preference.
  Interventions: Drug: Desloratadine; Drug: Zyrtec® (cetirizine)
- Zyrtec/RediTab (Active Comparator): Subjects received a single dose of Zyrtec chewable tablet followed 8-10 minutes later by a single dose of desloratadine RediTab followed thereafter by a statement of preference.
  Interventions: Drug: Desloratadine; Drug: Zyrtec® (cetirizine)

INTERVENTIONS:
Drug: Desloratadine — desloratadine RediTabs, 1 tablet (2.5 mg),oral administration, single day
  Other Names: SCH 034117
Drug: Zyrtec® (cetirizine) — Zyrtec® (cetirizine) Chewable Tablets, 1 tablet (5 mg), oral administration, single day

SUMMARY:
The primary objective of this study was to determine whether children ages 6-11 years prefer desloratadine RediTabs (2.5 mg) or a marketed competitor (Zyrtec® 5 mg Chewable Tablets). The secondary objectives of this study were to compare acceptance of the two attributes, taste and feeling in the mouth, of desloratadine 2.5 mg RediTabs and Zyrtec® 5 mg Chewable Tablets

ELIGIBILITY:
Inclusion Criteria:

* Subject and the parent/guardian of the subject, was to have demonstrated their willingness to participate in the study and comply with its procedures by signing a written Informed Consent
* 6-11 years old, either sex, either race
* If female, subject to be premenarcheal
* Willing to avoid eating, drinking, gum chewing, and teeth brushing for one hour prior to enrollment.
* Free of any clinically significant disease that would interfere with study evaluations, including allergic rhinitis and respiratory infections.
* Able to adhere to the dosing and visit schedules

Exclusion Criteria:

* If female, subject who was pregnant, intended to become pregnant during the study or nursing.
* Subject had used any investigational product within 30 days prior to enrollment.
* Subject had any of the following clinical conditions: history of any significant medical conditions (based on reporting by parent or guardian): e.g., diabetes, heart disease, liver disease, kidney disease, breathing problems, cough with excessive phlegm, or persistent or chronic cough.
* Subject had a current medical condition that, in the opinion of the Investigator or designee, may interfere with the ability to discriminate taste (e.g., common cold, sinus infection, bronchial infection, allergic rhinitis, etc.).
* Subject was participating in any other clinical study(ies).
* Subject was part of the staff or a family member of the staff personnel directly involved with this study.
* Subject was allergic to or has sensitivity to the study drug or its excipients.
* Subject had a history of allergic reaction to prescription and/or over the counter (OTC) medications and/or food products.
* Subject had used any antihistamines within 24 hours prior to tasting as outlined in Section 9.4.7.
* Subject used sedatives, tranquilizers, or monoamine oxidase inhibitor drugs.

Ages: 6 Years to 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 220 (Actual)
Dates: Start 2005-08; Primary Completion 2005-10 (Actual); Study Completion 2005-10 (Actual)

RESULTS

PARTICIPANT FLOW:
Groups:
- RediTab/Zyrtec: Subjects received a single dose of desloratadine Reditab followed 8-10 minutes later by a single dose of Zyrtec chewable tablet (first and second intervention period).
- Zyrtec/RediTab: Subjects received a single dose of Zyrtec chewable tablet followed 8-10 minutes later by a single dose of desloratadine RediTab (first and second intervention period).
Period: First Intervention
Arm/Group | RediTab/Zyrtec | Zyrtec/RediTab
Started | 109 | 111
Completed | 109 | 111
Not Completed | 0 | 0
Period: Interval Between Doses (8-10 Minutes)
Arm/Group | RediTab/Zyrtec | Zyrtec/RediTab
Started | 109 | 111
Completed | 109 | 111
Not Completed | 0 | 0
Period: Second Intervention
Arm/Group | RediTab/Zyrtec | Zyrtec/RediTab
Started | 109 | 111
Completed | 109 | 111
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total Population: All randomized subjects.
Arm/Group | Total Population
Number analyzed (Participants) | 220
Age, Continuous [Mean (Standard Deviation); unit: years] | 8.9 (1.65)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 109
  Male | 111

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects Who Preferred Desloratadine RediTab or Zyrtec Chewable Tablet.
Description: A product preference questionnaire was completed after the administration of the second study drug. An interviewer instructed the subject "now that you have tasted the two tablets, show us which tablet you like more" and the subject then marked which tablet he/she preferred. If the subject had no preference, the response was recorded accordingly.
Time Frame: Following the second dose (8-10 minutes after the first dose)
Population: All randomized subjects received either Reditab or Zyrtec, followed 8-10 minutes later by the opposite study drug (Reditab followed by Zyrtec or Zyrtec followed by Reditab).
Measure: Number; unit: participants
Groups:
- RediTab; Zyrtec; No Preference: All randomized subjects.
Arm/Group | RediTab | Zyrtec | No Preference
Number analyzed (Participants) | 220 | 220 | 220
participants | 149 | 33 | 38
Statistical Analysis 1: Comparison: RediTab vs Zyrtec; The Mainland-Gart test was applied to the preference rates in the subjects who showed a preference, to assess the difference in preference rates between RediTab and Zyrtec; Test type: Superiority or Other; p < 0.0001, Mainland-Gart Test — Statistical tests were performed at the significance level of 5%, without multiplicity adjustment; The p-value was derived from Mainland-Gart Test applied to a 2 (treatment sequence) by 2 (preferred period) contingency table

ADVERSE EVENTS:
Time Frame: 1 day
Arm/Group | RediTab/Zyrtec | Zyrtec/RediTab
Serious Adverse Events (participants affected / at risk) | 0/109 | 0/111
Other Adverse Events (participants affected / at risk) | 0/109 | 0/111

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The only disclosure restriction on the PI is that the sponsor can review results communications prior to release and can embargo communications regarding trial results for a period that is less than or equal to 45 days from the time submitted to the sponsor for review. If the parties disagree on the communication, the investigator and sponsor's representative will meet for the purpose of making a good faith effort to discuss and resolve any such issues or disagreement.